CLINICAL TRIAL: NCT00728819
Title: Peripherally Inserted Central Catheter (PICC) Thrombosis: Reverse Taper Versus Non-tapered Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 807264
Record Dates: First submitted 2008-07-31; First posted 2008-08-06 (Estimated); Results first posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-03

CONDITIONS: Venous Thrombosis
Keywords: Inpatients; Requiring; DL PICC; Access; Medications; Blood
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Tapered PICC
  Interventions: Device: Tapered PICC; Device: Non-tapered PICC
- 2 (Active Comparator): Non-tapered PICC
  Interventions: Device: Non-tapered PICC

INTERVENTIONS:
Device: Tapered PICC — Standard peripheral central catheter placement in the Brachial, Basilic or Cephalic veins
  Arms: 1
Device: Non-tapered PICC — Standard peripheral central catheter placement in the Brachial, Basilic or Cephalic veins

SUMMARY:
The purpose of this study is to compare two different marketed PICC (peripherally inserted central catheter) designs. Clotting rates, procedural bleeding and ease of catheter insertion will be compared. It is hypothesized that the non-tapered design has a lower clotting rate and is easier to place than the tapered design. Bleeding rates are expected to be about the same.

ELIGIBILITY:
Inclusion Criteria:

* All inpatients, age 18 to 90, in need of de novo central venous access with a double lumen catheter indication of > 2 weeks
* Informed consent and HIPAA consent forms discussed and signed by patient or their authorized representative

Exclusion Criteria:

* Skin related problems around the insertion site (infection, phlebitis, scars)
* History of mastectomy/axillary dissection on insertion side
* Coagulopathy with an INR of > 2.0
* Thrombocytopenia with platelets < 25,000 uL
* Renal insufficiency with a creatinine of > 3.0 mg/dL
* Documented current upper extremity or central venous thrombosis
* Hypercoagulable states (protein C or S deficiency, AT-III deficiency, lupus anticoagulant)
* Catheters needed for therapy within less than an hour (emergent placement not allowing sufficient time for proper research consent and randomization)
* Patient has already been enrolled in this research study
* Life expectancy less than 1 month

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2008-08; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Itkin, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Itkin M, Mondshein JI, Stavropoulos SW, Shlansky-Goldberg RD, Soulen MC, Trerotola SO. Peripherally inserted central catheter thrombosis--reverse tapered versus nontapered catheters: a randomized controlled study. J Vasc Interv Radiol. 2014 Jan;25(1):85-91.e1. doi: 10.1016/j.jvir.2013.10.009. Epub 2013 Nov 21. PMID 24268631

RESULTS

PARTICIPANT FLOW:
Groups:
- Taper PICC: Tapered PICC
  Tapered PICC: Standard peripheral central catheter placement in the Brachial, Basilic or Cephalic veins
  Non-tapered PICC: Standard peripheral central catheter placement in the Brachial, Basilic or Cephalic veins
- Non-tapered PICC: Non-tapered PICC
  Non-tapered PICC: Standard peripheral central catheter placement in the Brachial, Basilic or Cephalic veins
Period: Overall Study
Arm/Group | Taper PICC | Non-tapered PICC
Started | 171 | 168
Completed | 135 | 139
Not Completed | 36 | 29

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Taper PICC | Non-tapered PICC | Total
Number analyzed (Participants) | 171 | 168 | 339
Age, Customized [Count of Participants; unit: Participants]
  18-90 yo | 171 | 168 | 339
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 71 | 148
  Male | 94 | 97 | 191
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 171 | 168 | 339

OUTCOME MEASURES:

1. Primary Outcome: Evidence of PICC-related Venous Thrombosis
Description: Number participants with vein thrombosis
Time Frame: 28 days, PICC removal or hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Taper PICC | Non-tapered PICC
Number analyzed (Participants) | 139 | 135
Participants | 102 | 95

2. Secondary Outcome: Post-operative Bleeding
Description: Post-operative bleeding
Time Frame: Day 1
Population: Number of participants who received the intervention as assigned
Measure: Count of Participants; unit: Participants
Arm/Group | Taper PICC | Non-tapered PICC
Number analyzed (Participants) | 168 | 164
Participants | 4 | 9

3. Secondary Outcome: Symptomatic PICC-related Venous Thrombosis
Description: Symptomatic PICC-related venous thrombosis
Time Frame: Procedure through 28 days
Population: Number of participants who had this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Taper PICC | Non-tapered PICC
Number analyzed (Participants) | 167 | 164
Participants | 6 | 7

ADVERSE EVENTS:
Arm/Group | Taper PICC | Non-tapered PICC
Serious Adverse Events (participants affected / at risk) | 0/171 | 0/168
Other Adverse Events (participants affected / at risk) | 11/171 | 10/168
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taper PICC (N=171) | Non-tapered PICC (N=168)
Purelence (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
fever (Infections and infestations) | 10 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes